CLINICAL TRIAL: NCT03634176
Title: Optic Nerve Sheath Diameter in Retrobulbar Ultrasound as a Surrogate Measure for Intracranial Pressure Before and After Non-invasive Strategies
Status: Completed | Type: Observational
Sponsor: Hospital Dr. Miguel Pérez Carreño (Other)
Responsible Party: Principal Investigator, Aldo Saad Diab, Principal Investigator, anesthesiologist., Hospital Dr. Miguel Pérez Carreño
Other Study IDs: ABAY
Record Dates: First submitted 2018-08-11; First posted 2018-08-16 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Intracranial Hypertension; Optic Nerve Sheath Diameter
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group M: both optic nerve sheath diameter (the posterior 3mm of the papilla) before and after received 0.5gr/kg 20% mannitol
  Interventions: Diagnostic Test: optical nerve sheet diameter
- Group H: both optic nerve sheath diameter (the posterior 3mm of the papilla) before and after received 1.5 ml/kg 7.5% NaCl solution
  Interventions: Diagnostic Test: optical nerve sheet diameter
- Group P: both optic nerve sheath diameter (the posterior 3mm of the papilla) before and after patients were positioned on reverse Trendelenburg position 30 degrees higher than the feet
  Interventions: Diagnostic Test: optical nerve sheet diameter

INTERVENTIONS:
Diagnostic Test: optical nerve sheet diameter — The ONSD in each eye was measured vertically and horizontally 3 mm behind the optic disc, with the two values averaged. No pressure was applied to the orbit. At each time point, measurements were taken within 5 min. The measurements were made before (T1) and after some of the strategies according to group 30 min (T2), 60 min (T3), and 90 min (T4).

SUMMARY:
Measurement of the diameter of the sheath of the optic nerve in patients hospitalized in intensive care, with increased intracranial pressure (> 20mmHg) as a substitute measure for diagnosis and follow-up before and after different non-invasive strategies.

Three groups were created in which, through strategies already proven and non-invasive (mannitol, hypertonic solution 7.5% NaCl, reverse trendelenburg) to decrease the intracranial pressure, the optic nerve diameter measurement was performed and simultaneously the investigators monitored intracranial pressure through an intraventricular catheter continuously to determine if both correspond

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with traumatic or non-traumatic elevated ICP (defined as greater than 20 mm Hg for at least 10min)
* Hospitalized in ICU
* Patients with ICP continuous measurement through an intraventricular catheter
* Respiratory rate maintained at 10-18 breaths/min to maintain the end tidal carbon dioxide partial pressure between 35 and 40 mmHg
* Peak airway pressure <35 cmH2O
* Positive end-expiratory pressure <5 cmH2O

Exclusion Criteria:

* Patients who had undergone cranial decompression surgery
* Patients with ocular pathology
* Patients who had previously undergone eye surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit of the Dr. Migel Pérez Carreño hospital with increased intracranial pressure of traumatic or non-traumatic etiology.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheet diameter | immediately before administering the treatment according to the group and every 30 minutes after administering the treatment until 90 min.
  The optic nerve sheet diameter in each eye was measured vertically and horizontally 3 mm behind the optic disc, with the two values averaged

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dr Miguel Perez Carreño, Caracas, Venezuela, Bolivarian Republic of, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided